CLINICAL TRIAL: NCT02548520
Title: Vitamin D Status in the First 9 Months of Life
Brief Title: Maternal and Infant Vitamin Status During the First Nine Months of Infant Life
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: M-2007-0255
Record Dates: First submitted 2015-09-09; First posted 2015-09-14 (Estimated); Last update posted 2015-09-14 (Estimated); Status verified 2015-09

CONDITIONS: Rickets; Osteomalacia; Osteoporosis
MeSH Terms: conditions — Rickets; Osteomalacia; Osteoporosis | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Blood and breastmilk samples — The investigators collected maternal and infants blood samples from birth, and 4 and 9 months forward, including breastmilk from the mothers at all visits

SUMMARY:
In this study the investigators wanted to assess vitamin D status and possible consequences of low plasma 25-hydroxyvitamin D levels in a population of healthy mothers and their infants, in the community of Aarhus, Denmark.

DETAILED DESCRIPTION:
Danish people living at northern latitudes (56°N), often with overcast and foggy weather and few sunshine hours are at increased risk of vitamin D insufficiency. Although vitamin D is obtainable from fortified food and oily fish, the major source is the dermal synthesis of the vitamin D through exposure to solar ultraviolet light.

In the 19th century rickets was endemic in northern Europe, and many children developed rickets, a severe bone-deforming disease. Encouragement of sensible sun exposure, supplementation with cod liver oil and fortification of milk with vitamin D, resulted in an almost complete eradication of rickets by the end of the 19th century. At present vitamin D deficiency seems again to be more widespread. The classical outcomes of severe vitamin D deficiency are rickets in growing individuals and osteomalacia in adults. Low vitamin D status also relates to low bone density and increased risk of osteoporotic fractures. Although the incidence of rickets has declined over the last decades, cases attributable to inadequate vitamin D intake and low exposure to sunlight continue to be reported, and maternal vitamin D status may have permanent effects on newborns' health. Pregnant women, newborns, breastfed children, and lactating women are at a high risk of vitamin D deficiency, especially during winter and early spring.

Since fetal plasma 25-hydroxyvitamin D (25OHD) depends on maternal 25OHD, fetal vitamin D status may show seasonal changes parallel to those observed in the mothers. To prevent rickets and vitamin D deficiency in infants, most Western countries, including Denmark, recommend a daily maternal intake during pregnancy and lactation of 10 μg and that breastfed children are given a supplement of 10 μg of vitamin D/day. Despite these recommendations, approximately one third of Danish pregnant and lactating women have vitamin D insufficiency. However, childhood rickets is nowadays rare in Denmark, although it still exists especially among immigrants and mothers with prolonged lactation. Accordingly, in 2010, the Danish National Board of Health extended the recommendations for vitamin D supplementation to the first two years of life.

ELIGIBILITY:
Inclusion Criteria:

* Healthy pregnant Caucasian women aged 24-41 years,
* A normal pregnancy giving birth between 38-42 gestational weeks.

Exclusion Criteria:

* Chronic diseases,
* Other ethnic origin than Caucasian, and
* Alcohol or drug abuse.

Ages: 24 Years to 41 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy pregnant Caucasian women with a normal pregnancy
Sampling Method: Non-Probability Sample
Enrollment: 107 (Actual)
Dates: Start 2008-10; Primary Completion 2011-07 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Prevalence in plasma 25OHD and parathyroid hormone at birth | at birth (baseline)
  For determination of plasma 25OHD and plasma parathyroid hormone concentrations, the investigators sampled cord blood at baseline. Furthermore the investigators collected maternal blood at 2 weeks after birth (baseline).

SECONDARY OUTCOMES:
Prevalence in plasma 25OHD and parathyroid hormone at 4 months | at 4 months
  For determination of plasma 25OHD and plasma parathyroid hormone concentrations, the investigators sampled maternal and infants blood samples at 4 months (1. follow-up).
Prevalence in plasma 25OHD and parathyroid hormone at 9 months | at 9 months
  For determination of plasma 25OHD and plasma parathyroid hormone concentrations, the investigators sampled maternal and infants blood samples at 9 months (2. follow-up).

OTHER OUTCOMES:
Questionnaire about lifestyle factors at birth | at birth
  At birth the investigators collected, via self reported focused questionnaires, data regarding breastfeeding status, use of vitamin D supplements among children and their mothers, use of calcium supplements and dietary calcium intake (milk and cheese consumption) and other lifestyle factors, including physical activity (baseline).
Questionnaire about lifestyle factors at 4 months | at 4 months
  At 4 months the investigators collected, via self reported focused questionnaires, data regarding breastfeeding status, use of vitamin D supplements among children and their mothers, use of calcium supplements and dietary calcium intake (milk and cheese consumption) and other lifestyle factors, including physical activity (1. follow up).
Questionnaire about lifestyle factors at 9 months | at 9 months
  At 9 months visit the investigators collected, via self reported focused questionnaires, data regarding breastfeeding status, use of vitamin D supplements among children and their mothers, use of calcium supplements and dietary calcium intake (milk and cheese consumption) and other lifestyle factors, including physical activity (2. follow up).
peripheral Quantitative Computed Tomography i nine months old infants | at 9 months
  At 9 months the investigators investigated 1) whether there was a correlation between maternal vitamin D status or calcium intake (i.e. diet and supplements) and bone mass and structure as measured by peripheral quantitative computed tomography in the infants 9 months after birth, and 2) gender differences in measured peripheral quantitative computed tomography variables. Furthermore the investigators evaluated 3) the feasibility of performing peripheral quantitative computed tomography scans on newborn infants in terms of assessing the precision of peripheral quantitative computed tomography scan.

CONTACTS AND LOCATIONS:
Overall Officials: Susanna við Streym, PhD, Principal Investigator — Department of Internal Medicine and Endocrinology, Aarhus University Hospital; Lars Rejnmark, Professor, Study Director — Department of Internal Medicine and Endocrinology, Aarhus University Hospital; Peter Vestergaard, Professor, Study Chair — The Department of Endocrinology, Aalborg University Hospital
Locations (1):
- Department of Internal Medicine and Endocrinology, Aarhus University Hospital, Aarhus, Central Jutland, Denmark

REFERENCES:
- [Background] Vieth Streym S, Kristine Moller U, Rejnmark L, Heickendorff L, Mosekilde L, Vestergaard P. Maternal and infant vitamin D status during the first 9 months of infant life-a cohort study. Eur J Clin Nutr. 2013 Oct;67(10):1022-8. doi: 10.1038/ejcn.2013.152. Epub 2013 Sep 4. PMID 24002039
- [Derived] vieth Streym S, Hojskov CS, Moller UK, Heickendorff L, Vestergaard P, Mosekilde L, Rejnmark L. Vitamin D content in human breast milk: a 9-mo follow-up study. Am J Clin Nutr. 2016 Jan;103(1):107-14. doi: 10.3945/ajcn.115.115105. Epub 2015 Dec 16. PMID 26675779